CLINICAL TRIAL: NCT06325007
Title: The Effect of Combining Single Balloon Catheter With Castor Oil Ingestion for Cervical Ripening on Time to Delivery Among Nulliparous Women.
Brief Title: Castor Oil Ingestion and Balloon Catheter for Labor Induction in Nulliparous
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holy Family Hospital, Nazareth, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, head of obstetrics and gynecology department, Holy Family Hospital, Nazareth, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 293-2024-HFH
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 - study group (Active Comparator): Candidates will drink a mixture of 60 ml of castor oil and 140 ml of orange juice. 30 minutes later, A 22-French Foley catheter will be inserted above internal cervical os and will be filled with 60 mL of normal saline.
  Interventions: Dietary Supplement: Induction of labor
- group 2- control (Active Comparator): A foley catheter will be inserted into cervical canal as described above according to the department protocol without ingestion of castor oil.
  Interventions: Dietary Supplement: Induction of labor

INTERVENTIONS:
Dietary Supplement: Induction of labor — The study group only will drink a mixture of 60 ml of castor oil mixed with 140 ml of orange juice. Thirty minutes later, in both groups, an extraamniotic single balloon catheter will be inserted above the internal cervical os and filled with 60 mL of normal saline. Following removal, artificial rupture of the membranes will be performed as long as it is safe with regards to fetal head position. Oxytocin infusion will be commenced at once if contraction has not begun spontaneously (2 to 3 regular uterine contractions per 10 minutes). Continuous electronic fetal monitoring will be used throughout labor. Labor will be managed by the attending obstetricians and midwives. Labor progress abnormalities will be diagnosed and managed according to the department protocol based on the recommendations of the American College of Obstetricians and Gynecologists.

SUMMARY:
The goal of this randomized controlled trial is to examine the efficacy of combining castor oil ingestion with extra-amniotic single balloon catheter for cervical ripening on time from induction to delivery in nulliparous women.

The main question it aims to answer are:

Does the addition of the use of castor oil to extra-amniotic single balloon reduce the time until birth? Does the addition of the castor oil affect other perinatal outcomes during childbirth? Are the side effects of the castor tolerated by the mothers? Participants will be randomly divided into 2 groups: the study group will drink a mixture of 60 ml of castor oil mixed with 140 ml of orange juice. Thirty minutes later, an extra-amniotic single balloon catheter will be inserted above the internal cervical os and filled with 60 mL of normal saline. In the control group, a foley catheter will be inserted into cervical canal without ingestion of castor oil.

DETAILED DESCRIPTION:
The rate of labor induction has increased up to 25.7% in 2018 for several demographic and obstetric reasons. In nulliparous women the reported rate is nearly 32%.

Various methods are used to induce labor worldwide, including natural, mechanical and pharmacological agents. of all methods balloon catheters were proven to cause fewer adverse perinatal events.

Though induction is considered a safe and effective procedure, it may lead to a prolonged labor which is associated with complications such postpartum hemorrhage, infection, and operative delivery.

Based on these data several studies have examined the combinations of balloon catheters with other pharmacological agents on labor durations. The results were inconsistent, and several reports showed that the combination reduced significantly the length of labor. Nevertheless, pharmacological agents may be associated with adverse events including uterine hyperstimulation, placental abruption, and postpartum hemorrhage, though the overall risk is small.

Castor oil, extracted from the seeds of Ricinus communis plant, is a natural effective substance for induction of labor. it's considered a safe and inexpensive though the exact mechanism by which it induces labor is still unclear.

Our hypothesis suggests that ingestion of castor oil combined with the balloon catheter will shorten the time to delivery. In order to show a reduction by 3 hours, a sample size of 57 in each group will be needed assuming 80% power and a two-tailed alpha of 5%.

Since the success rate of vaginal delivery is nearly 85%, the sample size was calculated to 67 women in each group. Additional 5% are planned to be recruited to account for trial drop out for any reason, yielding a total final sample size of 71 women in each group (142 in both groups).

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years old
* Sign an informed consent
* Term pregnancy (>37 weeks)
* Viable fetus
* Singleton
* Vertex presentation
* Intact membranes
* Cervix with Bishop score ≤6

Exclusion Criteria:

* Previous cesarean delivery
* Major fetal malformations
* Contraindication to spontaneous vaginal delivery
* Amniotic fluid index >25cm
* Chorioamnionitis at admission
* Placental abruption
* Previous prostaglandin use for induction of labor
* A low-lying placenta (up to 2 cm from the internal os)
* Carriers of hepatitis B or C or human immunodeficiency viruses
* Women with a history of allergy to latex.
* Women with a history of allergy to castor oil

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 142 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
time to delivery | 48 hours
  Time from catheter insertion to vaginal delivery.

SECONDARY OUTCOMES:
balloon expulsion time | 12 hours after insertion
  The time until balloon was spontaneously expelled
Bishop score after catheter expulsion | 12 hours
  Bishop score after removal of the catheter where a high score (above 7) indicates a better outcome.
Fetal presentation at the delivery | 48 hours
  The insertion of a balloon may lead to a change in the presenting part of the fetus. A change to a non-vertex presentation is carried as an undesired outcome.
Duration of the active phase of labor | 4 hours
  Duration of the time from 6 cm cervical dilatation to 10 cm cervical dilatation
Duration of second stage | 4 hours
  the time from 10 cm cervical dilatation until the delivery of the baby
Mode of delivery | 48 hours
  Whether the birth was a normal spontaneous birth, operative vaginal birth or a cesarean section.
Indications for cesarean or operative vaginal deliveries | 48 hours
  Was the reason for operative vaginal delivery or cesarean delivery due to non progress labor, fetal status, or a combination of both?
Intrapartum fever | 48 hours
  Number of patients that will have intrapartum fever ≥ 38 °C
Number of patients that will require use of intrapartum use of antibiotic treatment. | 48 hours
  Number of patients that will require use of intrapartum use of antibiotic treatment due to intrapartum infection.
Number of Participants with that will develop clinical signs of chorioamnionitis. | 48 hours
  Clinical signs of chorioamnionitis includes abdominal tenderness, abnormal discharge, intrapartum fever, tachycardia
Number of Participants with that will develop 3rd and 4th degrees perineal lacerations. | 48 hours
  Obstetric anal sphincter injury
Number of Participants with develop postpartrum hemorrhage. | 48 hours
  early postpartum hemorrhage (PPH)
Number of Participants with need blood transfusion. | 72 hours
  PPH that required blood transfusion
Side effects related to castor oil use | 48 hours
  nausea, vomiting, uterine hyperstimulation> the 5 contractions: 10 minutes
Oxytocin maximal dosage | 48 hours
  Oxytocin maximal dosage
Number of participants with Umbilical Cord prolapse. | 48 hours
  Umbilical cord prolapse is when the umbilical cord exits the cervical os before the fetal presenting part that may result in fetal hypoxia.
Apgar score (0 to 10). | 48 hours
  APGAR< 7 after 1 and 5 minutes where lower scores mean a worse outcome.
pH taken from umbilical artery | 48 hours
  Cord artery pH <7.1
Neonatal birthweight | 48 hours
  Neonatal birthweight
Number of neonates with Neonatal fever ≥ 38 °C | 72 hours
  Neonatal fever >38
The number of neonates that will develop neonatal sepsis. | 72 hours
  Diagnosis of neonatal sepsis based on clinical signs of sepsis and positive cultures.
The number of neonates that will require antibiotic treatment. | 72 hours
  Need for antibiotic treatment
Neonatal complications | 48 hours
  respiratory distress syndrome, transient tachypnea of newborn, intracranial hemorrhage, intraventricular hemorrhage, seizures, Meconium aspiration syndrome ,Hypoxic ischemic encephalopathy
The number of neonates that will Admit to neonatal intensive care unit (NICU) | 30 days
  Neonatal admission to NICU
Length of stay in NICU. | 30 days
  Neonatal length of stay in NICU.
neonatal death | 30 days
  neonatal death
Maternal hemoglobin level after delivery. | 48 hours
  higher level of Hemoglobin and indicate better outcome.
Number of participants that will require postpartum hysterectomy. | 72 hours following delivery.
  Maternal hysterectomy
Number of participants that will require postpartum laparotomy. | 72 hours following delivery.
  Number of participants that will require postpartum laparotomy after vaginal delivery or re-laparotomy after cesarean section.
postpartum maternal complications | 72 hours following the delivery.
  endometritis
The length of stay from birth to discharge home. | up to 10 days
  The length of stay in days from birth to discharge home.
Maternal satisfaction from delivery process. | up to 10 days after delivery
  1 = Very dissatisfied, 10 = Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — Holy Family Hospital, Nazareth, Israel
Locations (2):
- Israel (2):
  - Holy Family hospital, Nazareth, Nazareth
  - Holy Family Hospital, Nazareth

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Access to IPD can be requested by qualified researchers and will be granted after review and approval of a research proposal and statistical analysis plan and execution of a data sharing agreement. For more information or to apply, please contact the Principal Investigator

REFERENCES:
- [Result] 1.Clinical management guidelines for Obstetrician-Gynecologists. The American College of Obstetricians and Gynecologists 2009. Vol.114, No.2, Part1. 2. Grobman W, et al. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. The new England journal of medicine 2018;379;6. 3. Jones MN,et al. Balloon catheters versus vaginal prostaglandins for labour induction (CPI Collaborative): an individual participant data meta-analysis of randomised controlled trials. Lancet 2022;400:1681-1692. 4. Cheng YW, et al. The association between the length of first stage of labor, mode of delivery, and perinatal outcomes in women undergoing induction of labor. Am J Obstet Gynecol. 2009;201:477.e1-7. 5. Cheng YW, et al. Length of the first stage of labor and associated perinatal outcomes in nulliparous women. Obstet Gynecol 2010;116:1127-35. 6. Gagnon J, et al. Intracervical Foley catheter with and without oxytocin for labor induction with Bishop score ≤3: a secondary analysis. Am J Obstet Gynecol MFM 2021;3:100350. 7. Edwards RK, et al. Controlled Release Dinoprostone Insert and Foley Compared to Foley Alone: A Randomized Pilot Trial. Am J Perinatol 2021;38:e57-e63. 8. DeMariaa A, et al. Castor oil as a natural alternative to labor induction: A retrospective descriptive study. Women and Birth 2018;31:e99-e104. 9. Moradi M, et al. Effect of Castor Oil on Cervical Ripening and Labor Induction: a systematic review and meta-analysis. Journal Of Pharmacopuncture 2022;25:71-78. 10. Shalev-Ram H, et al. Is there a difference in labor patterns after induction with prostaglandins and double-balloon catheters? American Journal of Obstetrics and Gynecology 2023;3:100198. 11. Tunarua S, et al. Castor oil induces laxation and uterus contraction via ricinoleic acid activating prostaglandin EP3 receptors. Proceedings of the National Academy of Sciences 2012. 12. Kelly AJ, et al. Castor oil, bath and/or enema for cervical priming and induction of labour. Cochrane Database Syst Rev 2013;2013:CD003099. 13. Bayoumi YA, et al. Castor oil for labor initiation in women with a previous cesarean section: a double-blind randomized study. J Matern Fetal Neonatal Med 2022;35:8945-8951. 14. Gilada R, et al. Castor oil for induction of labor in post-date pregnancies: A randomized controlled trial. Women and Birth 2018;e26-e31. 15. Salim R, et al. Single-balloon compared with double-balloon catheters for induction of labor: a randomized controlled trial. Obstet Gynecol 2011;118:79-86. 16. American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, et al. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol 2014;210:179-93.